CLINICAL TRIAL: NCT03952091
Title: A Phase 3, Randomized, Open-label, Parallel-controlled, Multi-center Study Comparing TJ202, Lenalidomide and Dexamethasone vs. Lenalidomide and Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma Who Received at Least 1 Prior Line of Treatment
Brief Title: TJ202, Lenalidomide and Dexamethasone vs. Lenalidomide and Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ202001MMY301
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma in Relapse; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TJ202, Lenalidomide and Dexamethasone (Experimental)
  Interventions: Drug: TJ202, Lenalidomide and Dexamethasone
- Lenalidomide and Dexamethasone (Active Comparator)
  Interventions: Drug: Lenalidomide and Dexamethasone

INTERVENTIONS:
Drug: TJ202, Lenalidomide and Dexamethasone — One dose of TJ202 will be given on Day 1 and Day 4 of Week 1, respectively, every week from Week 2 to Week 12, every 2 weeks from Week 13 to Week 24 and then every 4 weeks thereafter.Lenalidomide 25mg will be administered orally on Days 1 through 21 of each 28-days cycle.Dexamethasone 40 mg will be administered on Day 1 and Day 4 of Week 1, respectively and then 40mg weekly thereafter.
  Arms: TJ202, Lenalidomide and Dexamethasone
Drug: Lenalidomide and Dexamethasone — Lenalidomide 25mg will be administered orally on Days 1 through 21 of each 28-days cycle.Dexamethasone 40 mg weekly will be administered.
  Arms: Lenalidomide and Dexamethasone

SUMMARY:
A phase 3, randomized, open-label, parallel-controlled, multi-center study comparing TJ202, Lenalidomide and Dexamethasone vs. Lenalidomide and Dexamethasone in subjects with relapsed or refractory multiple myeloma who received at least 1 prior line of treatment

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18, male or female;
2. Subjects must have had documented MM;
3. At the screening phase, subject must have one or more measurable disease;
4. Subjects must have received at least 1 prior line treatment* for relapsed or refractor MM;
5. Subjects who are in a state of progressive disease (PD);
6. Subjects must have life expectancy of no less than 6 months;
7. Subjects must have an ECOG (Eastern Cooperative Oncology Group) performance status score of 0~2;
8. A woman of child-bearing potential must have a negative serum pregnancy test within 14 days prior to the first study agent administration, and a negative urine pregnancy test on the day of the first study agent administration; as well as those should avoid sexual intercourse with the opposite sex or should adopt two reliable methods of contraception at the same time during the study period. A woman of child-bearing potential is required to take effective contraceptive measures throughout this study and within 6 months after the last dosing; female subjects must agree not to donate any eggs for the purpose of assisted reproduction throughout this study and within 6 months after completion of this study;
9. Male subjects who are sexually active with women of child-bearing potential and have not undergone vasoligation must agree to use barrier methods of birth control, or that their partners use block caps (cervical cap or dome cap), spermicidal foam, contraceptive gel, contraceptive diaphragm, contraceptive cream, or suppository, and all male subjects are not allowed to donate sperms throughout this study and within 6 months after the last dosing;
10. Subject must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study;
11. Subject must be willing and able to adhere to the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

1. Subject has received anti-CD38 monoclonal antibody treatment previously;
2. Subject has received CAR-T cell therapy previously;
3. Subject has previously received allogenic stem cell transplant, or subject has received autologous stem cell transplant within 3 months before administration of the study agent;
4. Primary refractory multiple myeloma;
5. Subject's disease shows evidence of resistance to lenalidomide;
6. Subject's disease shows evidence of intolerance to lenalidomide;
7. Subject is exhibiting clinical signs of central nervous system (CNS) involvement of MM;
8. Subjects with known moderate or severe persistent asthma within the past 5 years;
9. Subject has active hepatitis B or C virus infection15. Subject is seropositive for human immunodeficiency virus (HIV);
10. Subject has clinically significant cardiac disease;
11. Subject has known allergies, hypersensitivity, or intolerance to lenalidomide, corticosteroids, monoclonal antibodies or human proteins, or their excipients or known sensitivity to mammalian-derived products;
12. Subject with known or suspicious conditions that would lead to failure to abide by the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 18.4 months(Active) 30.7 months(experimental)
  defined as the duration from the date of randomization to either PD, according to the IMWG criteria, or death, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (39):
- China (38):
  - Capital Medical University (CMU) - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Bengbu Medical college, Bengbu, Bengbu
  - The First Bethune Hospital of Jilin University, Jilin, Changchun
  - Hunan Cancer Hospital, Hunan, Changsha
  - Fujian Medical University Union Hospital, Fujian, Fuzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center, Guangdong, Guangzhou
  - Guangdong General Hospital, Guangdong, Guangzhou
  - Guangzhou First People's Hospital, Guangdong, Guangzhou
  - Nanfang Hospital, Guangdong, Guangzhou
  - The First Affiliated Hospital of Zhejiang University, Zhejiang, Hangzhou
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Chang Gung Medical Foundation - Kaohsiung Chang Gung Memorial Hospital, Taiwan, Kaohsiung
  - The second affiliated hospital of Kunming medical university, Yunnan, Kunming
  - The First People's Hospital of Yunnan Province, Yunnan, Kunming
  - The First Hospital of Lanzhou University, Lanzhou, Lanzhou
  - Lanzhou University Second Hospital, Lanzhou, Lanzhou
  - Second Affiliated Hospital of Nanchang University, Jiangxi, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing, Nanjing
  - Jiangsu Province Hospital, Nanjing, Nanjing
  - Guangxi Medical Univ. 1st Hospital, Guangxi, Nanning
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Shanghai Jiao Tong University School of Medicine - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - The First Hospital of China Medical University, Shenyang, Shenyang
  - Shenzhen Second Hospital, Guangdong, Shenzhen
  - The First Affiliated Hospital of Soochow University, Suzhou, Suzhou
  - National Taiwan University Hospital, Taiwan, Taibei
  - Taichung Veterans General Hospital, Taiwan, Taichung
  - Tri-Service General Hospital, Taiwan, Taipei
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Wenzhou Medical University, Zhejiang, Wenzhou
  - The Central Hospital Of Wuhan, Hubei, Wuhan
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Henan Cancer Hospital, Henan, Zhengzhou
- Taipei Veterans General Hospital, Taipei, Taiwan